CLINICAL TRIAL: NCT00496977
Title: Screening for Lung Cancer. A Randomised Controlled Trial of Low-Dose CT-Scanning.
Brief Title: Danish Lung Cancer Screening Trial (DLCST)
Acronym: DLCST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danish Lung Cancer Group (Other)
Collaborators: Ministry of the Interior and Health, Denmark (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: KA-02045
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-06

CONDITIONS: Lung Cancer
Keywords: lung cancer; CT scan; screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: annual CT screening

SUMMARY:
The trial is a randomised trial comparing annual CT screening for lung cancer with no screening in 4104 smokers and former smokers between the age of 50 and 70 years. The goals are: 1) to evaluate if annual CT screening can reduce lung cancer mortality by more than 20 % (in collaboration with the NELSON trial in the Netherlands, 2) to evaluate psychological effects of screening including the effects of false positive diagnoses, and 3) to evaluate possible effects on smoking behaviour. The trial is funded in full by the Danish Ministry of Interior and Health.

DETAILED DESCRIPTION:
The trial is a parallel randomized controlled trial comparing either a yearly low dose CT scan or no screening. It is scheduled to enroll 4000 smokers and former smokers, and the study is scheduled to last 5 years, i.e. an initial (prevalence) screening is followed by 4 annual (incidence) screenings.

In addition the following investigations are done: A prospective, longitudinal questionnaire assessment of enrolled participants who have received a false positive diagnosis. The questionnaire will focus on the consequences of receiving a false positive diagnosis. Answers from enrolled subjects who have received a false positive diagnosis will be compared to their own "baseline" responses, and responses from subjects who have received a negative result of their own low-dose CT scans All participants will annually be questioned regarding smoking habits, their motivation for cessation of smoking and will be advised to refrain from smoking to assess the effect of participation in a screening protocol for lung cancer on cessation of smoking.

Socioeconomic consequences of screening for lung cancer will be assessed by longitudinal registration of costs and benefits (e.g. morbidity, hospitalization, GP consultations etc.

Assess the value of PET scanning when screening for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Smoking exposure > 20 pack years
* Quit smoking < 10 years
* Fit to undergo treatment
* Pulmonary function test > 30 % of expected (FEV1)

Exclusion Criteria:

* Bodyweight > 130 Kg
* Formely treated for lungcancer, breastcancer, melanoma or hypernephroma.
* Serious co-morbidity with life expectancy below 10 years.
* Treated for other malignant diseases within the last 5 years.
* Treatment for pulmonary tuberculosis within the last 2 years.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4104 (Actual)
Dates: Start 2004-10; Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Lung cancer mortality | 10 years

SECONDARY OUTCOMES:
lung cancer incidense and stagedistribution | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jesper H Pedersen, MD, Dr.Sci, Principal Investigator — Gentofte University Hospital, Hellerup, Denmark
Locations (1):
- Lung Screening Clinic, Gentofte University Hospital, Hellerup, Denmark

REFERENCES:
- [Derived] Venkadesh KV, Aleef TA, Scholten ET, Saghir Z, Silva M, Sverzellati N, Pastorino U, van Ginneken B, Prokop M, Jacobs C. Prior CT Improves Deep Learning for Malignancy Risk Estimation of Screening-detected Pulmonary Nodules. Radiology. 2023 Aug;308(2):e223308. doi: 10.1148/radiol.223308. PMID 37526548
- [Derived] Rasmussen JF, Siersma V, Malmqvist J, Brodersen J. Psychosocial consequences of false positives in the Danish Lung Cancer CT Screening Trial: a nested matched cohort study. BMJ Open. 2020 Jun 4;10(6):e034682. doi: 10.1136/bmjopen-2019-034682. PMID 32503869
- [Derived] Malmqvist J, Siersma V, Thorsen H, Heleno B, Rasmussen JF, Brodersen J. Did psychosocial status, sociodemographics and smoking status affect non-attendance in control participants in the Danish Lung Cancer Screening Trial? A nested observational study. BMJ Open. 2020 Feb 20;10(2):e030871. doi: 10.1136/bmjopen-2019-030871. PMID 32086352
- [Derived] Jensen MD, Siersma V, Rasmussen JF, Brodersen J. Direct and indirect healthcare costs of lung cancer CT screening in Denmark: a registry study. BMJ Open. 2020 Jan 21;10(1):e031768. doi: 10.1136/bmjopen-2019-031768. PMID 31969362
- [Derived] Wille MM, Dirksen A, Ashraf H, Saghir Z, Bach KS, Brodersen J, Clementsen PF, Hansen H, Larsen KR, Mortensen J, Rasmussen JF, Seersholm N, Skov BG, Thomsen LH, Tonnesen P, Pedersen JH. Results of the Randomized Danish Lung Cancer Screening Trial with Focus on High-Risk Profiling. Am J Respir Crit Care Med. 2016 Mar 1;193(5):542-51. doi: 10.1164/rccm.201505-1040OC. PMID 26485620
- [Derived] Winkler Wille MM, van Riel SJ, Saghir Z, Dirksen A, Pedersen JH, Jacobs C, Thomsen LH, Scholten ET, Skovgaard LT, van Ginneken B. Predictive Accuracy of the PanCan Lung Cancer Risk Prediction Model -External Validation based on CT from the Danish Lung Cancer Screening Trial. Eur Radiol. 2015 Oct;25(10):3093-9. doi: 10.1007/s00330-015-3689-0. Epub 2015 Mar 13. PMID 25764091
- [Derived] Rasmussen JF, Siersma V, Pedersen JH, Brodersen J. Psychosocial consequences in the Danish randomised controlled lung cancer screening trial (DLCST). Lung Cancer. 2015 Jan;87(1):65-72. doi: 10.1016/j.lungcan.2014.11.003. Epub 2014 Nov 20. PMID 25433982
- [Derived] Ashraf H, Saghir Z, Dirksen A, Pedersen JH, Thomsen LH, Dossing M, Tonnesen P. Smoking habits in the randomised Danish Lung Cancer Screening Trial with low-dose CT: final results after a 5-year screening programme. Thorax. 2014 Jun;69(6):574-9. doi: 10.1136/thoraxjnl-2013-203849. Epub 2014 Jan 17. PMID 24443174
- [Derived] Thomsen LH, Dirksen A, Shaker SB, Skovgaard LT, Dahlback M, Pedersen JH. Analysis of FEV1 decline in relatively healthy heavy smokers: implications of expressing changes in FEV1 in relative terms. COPD. 2014 Feb;11(1):96-104. doi: 10.3109/15412555.2013.830096. Epub 2013 Oct 10. PMID 24111638
- [Derived] Rasmussen T, Frestad D, Kober L, Pedersen JH, Thomsen LH, Dirksen A, Kofoed KF. Development and progression of coronary artery calcification in long-term smokers: adverse effects of continued smoking. J Am Coll Cardiol. 2013 Jul 16;62(3):255-257. doi: 10.1016/j.jacc.2013.04.013. Epub 2013 Apr 30. No abstract available. PMID 23643591
- [Derived] Kaerlev L, Iachina M, Pedersen JH, Green A, Norgard BM. CT-Screening for lung cancer does not increase the use of anxiolytic or antidepressant medication. BMC Cancer. 2012 May 23;12:188. doi: 10.1186/1471-2407-12-188. PMID 22621716
- [Derived] Saghir Z, Ashraf H, Dirksen A, Brodersen J, Pedersen JH. Contamination during 4 years of annual CT screening in the Danish Lung Cancer Screening Trial (DLCST). Lung Cancer. 2011 Mar;71(3):323-7. doi: 10.1016/j.lungcan.2010.06.006. PMID 20619924